CLINICAL TRIAL: NCT02112526
Title: An Open-label, Phase 1b Study of ACP 196 in Subjects With Relapsed or Refractory de Novo Activated B-cell (ABC) Subtype of Diffuse Large B-Cell Lymphoma
Brief Title: Acalabrutinib (ACP-196), a Btk Inhibitor, for Treatment of de Novo Activated B-cell (ABC) Subtype of Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-002; 2014-001341-25 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Activated B-cell Diffuse Large B-Cell Lymphoma (ABC DLBCL)
Keywords: de Novo Activated B-cell (ABC) Subtype of Diffuse Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma; de Novo Activated B-cell (ABC); de Novo Activated B-cell; ABC DLBCL; DLBCL; Lymphoma; B-Cell; Immunoproliferative Disorders; Immune System Diseases; Bruton's tyrosine kinase
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Immunoproliferative Disorders; Immune System Diseases | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acalabrutinib (Experimental)
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib
  Other Names: ACP-196

SUMMARY:
To characterize the safety profile of acalabrutinib in subjects with relapsed or refractory de Novo Activated B-cell (ABC) Subtype of Diffuse Large B-Cell Lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Pathologically confirmed de novo ABC DLBCL
* Relapsed or refractory disease
* Subjects must have ≥ 1 measurable disease sites

Exclusion Criteria:

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or LVEF < 50%
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Breast feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Clinical Trials, Study Director — 1-877-240-9479; information.center@astrazeneca.com
Locations (7):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Atlanta, Georgia
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Houston, Texas
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  htttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  URL:
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-002&attachmentIdentifier=a4c264ed-fa39-4838-ab81-34e825c02b50&fileName=ACE-LY-002_Protocol_Amendment_V4_dated_16Mar2020-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-002&attachmentIdentifier=679c0d48-ae9f-49dd-af1f-a404914a80d9&fileName=ACE-LY-002_Final_Safety_Report_CSR_Synopsis_Ed_2_dated_14Nov2018-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Relapse Subjects; Cohort 2 - Refractory Subjects: Acalabrutinib 100mg administered orally (PO) twice daily (BID)
Period: Overall Study
Arm/Group | Cohort 1 - Relapse Subjects | Cohort 2 - Refractory Subjects
Started | 11 | 10
Enrolled | 11 | 10
Received Study Medication | 11 | 10
Discontinued Study | 11 | 9
Subjects Continuing Study Medication | 0 | 1
Completed | 0 | 1
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Relapse Subjects | Cohort 2 - Refractory Subjects | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: Year] | 70.7 (9.57) | 56.9 (16.26) | 64.1 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 6 | 15
  United Kingdom | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Acalabrutinib in Subjects With Relapsed or Refractory ABC DLBCL.
Description: Safety assessments included SAEs TEAEs, including AEs leading to discontinuation of study drug or dose reduction.
Time Frame: SAEs collected from time of consent; TEAEs beginning after first dose and continuing through 30 days (+/- 7 days) after last dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Relapse Subjects | Cohort 2 - Refractory Subjects
Number analyzed (Participants) | 11 | 10
Participants | 3 | 2

2. Secondary Outcome: Area Under the Plasma Concentration (AUC)
Description: To Characterize the Pharmacokinetic parameter AUC of acalabrutinib
Time Frame: 1 Cycle (28 days)
Reporting Status: Not Posted

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: To Characterize the Pharmacokinetic parameter Cmax of acalabrutinib
Time Frame: 1 Cycle (28 days)
Reporting Status: Not Posted

4. Secondary Outcome: Evaluate Pharmacodynamic (PD) Effects (Done at US Sites Only)
Description: To evaluate the concentration pharmacodynamic effects of acalabrutinib
Time Frame: 2 Cycles (1 cycle = 28 days) and at end of treatment
Reporting Status: Not Posted

5. Secondary Outcome: Evaluate Activity of Acalabrutinib as Measured by Overall Response Rate (ORR)
Description: To evaluate the activity of acalabrutinib as measured by ORR
Time Frame: From enrollment to the date of disease progression, assessed up to Cycle 48 (1 cycle is 28 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and on or before Day 697
Groups:
- Cohort 1 - Relapse Subjects; Cohort 2 - Refractory Subjects: Acalabrutinib 100mg administered orally (PO) twice daily
Arm/Group | Cohort 1 - Relapse Subjects | Cohort 2 - Refractory Subjects
All-Cause Mortality (participants affected / at risk) | 3/11 | 5/10
Serious Adverse Events (participants affected / at risk) | 4/11 | 5/10
Other Adverse Events (participants affected / at risk) | 10/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Relapse Subjects (N=11) | Cohort 2 - Refractory Subjects (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Influenza B virus test positive (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Relapse Subjects (N=11) | Cohort 2 - Refractory Subjects (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4
Oedema peripheral (General disorders) | 2 | 2
Gait disturbance (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Axillary pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Injection site bruising (General disorders) | 1 | 0
Injection site rash (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 3 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Urinary retention disorders (Renal and urinary disorders) | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02112526/Prot_004.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02112526/SAP_001.pdf